CLINICAL TRIAL: NCT04575428
Title: Splanchnic Nerve Block for Therapy of Chronic Heart Failure (Splanchnic III)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103788
Record Dates: First submitted 2020-08-20; First posted 2020-10-05 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Chronic Heart Failure
Keywords: heart failure, exercise, splanchnic nerve block
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Splanchnic nerve block (Experimental)
  Interventions: Drug: Splanchnic nerve block

INTERVENTIONS:
Drug: Splanchnic nerve block — Percutaneous splanchnic nerve block

SUMMARY:
Splanchnic vasoconstriction may contribute to decompensation of chronic heart failure (HF) via volume redistribution from the splanchnic vascular bed to the central compartment. This is a sympathetically mediated reflex and can be interrupted through a splanchnic nerve block (SNB). We hypothesize that interruption of the efferent/afferent innervation of the splanchnic vasculature will decrease cardiac congestion in patients presenting with HF. Based on preliminary safety and efficacy data in acute and chronic heart failure patients with temporary (<24 h) SNB. Now we will apply a prolonged SNB in chronic heart failure patients using a long acting agent. We will test the effects of SNB on long term exercise capacitance.

DETAILED DESCRIPTION:
Activation of splanchnic nerves results in vasoconstriction and reduces splanchnic capacitance, therefore recruiting blood volume into the central circulation. In heart failure, a reduced splanchnic vascular capacitance could be the mechanism underlying symptoms of exercise intolerance and could predispose to rapid decompensation with external fluid intake or retention. A compromised vascular reservoir is likely unable to buffer shifts of fluid and actively contributes to the acute or chronic expulsion of fluid from the splanchnic vascular compartment to the central thoracic compartment. The redistribution of blood volume into the central circulation may lead to a sudden rise in pulmonary and left-sided cardiac pressures in HF. This makes the splanchnic vascular compartment an attractive target in heart failure. Our preliminary proof-of-concept work in patients with acute decompensated and chronic heart failure showed promise for the concept of splanchnic nerve modulation in heart failure. In a series of two small first-in-human studies for acute decompensated heart failure (N=13) (NCT02669407) and chronic heart failure (N=17) (NCT03453151), we found that a splanchnic nerve block (SNB) with lidocaine (90 min duration of action) and ropivacaine (24 hours duration of action) acutely reduced resting and exercise-induced intra-cardiac filling pressures, associated with improved patient symptoms and functional capacity.

The present study will be a prospective open-label pilot study to help establish feasibility, safety and enable dose finding for botulinumtoxin. Following a baseline invasive (right heart catheterization) cardiopulmonary exercise testing (CPX) patients will undergo unilateral celiac plexus block, followed by repeat hemodynamic testing. Functional testing at baseline and follow up will be supplemented by measures of blood volume and autonomic tone.

ELIGIBILITY:
Inclusion Criteria:

* Followed at DUMC for known or suspected diagnosis of HF (NYHA stage 2-4, Class C-D), including patients on inotropic medication
* Systolic blood pressure (SBP) > 100 mmHg
* History of HF hospitalization or ER visit or iv diuretic use in last 12 months.
* Patients will be included regardless of left ventricular ejection fraction.

Exclusion Criteria:

* Anticoagulation at the time the procedure or in case of recent warfarin use an INR >1.4. Anticoagulation includes: warfarin, or novel oral anticoagulants like dabigatran, rivaroxaban, apixaban, endoxaban or full dose intravenous heparin products or bivalirudin and fondaparinux). Antiplatelet agents besides aspirin such as ticagrelor, prasugrel, Plavix are also considered to be a contraindication if used at time point of procedure.
* Immunosuppressive medications for solid organ transplant
* Acute MI (STEMI or Type I NSTEMI) within 7 days?
* Evidence of progressive cardiogenic shock within 48 hours
* Restrictive cardiomyopathy
* Constrictive pericarditis
* Pericardial effusion with evidence of tamponade
* Severe valvular stenosis requiring intervention
* Known history of an increased bleeding risk
* Thrombocytopenia (< 50,000)
* End-stage renal disease CKD stage 5 due to primary renal pathology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marat Fudim, MD, MHS, Principal Investigator — Duke Universtiy
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Splanchnic Nerve Block
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Left ventricular ejection fraction >55% [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Peak Exercise Wedge Pressure
Description: Measured with cardiopulmonary exercise testing
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Mmhg
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
Mmhg
  Pre nerve block | 44 (6.2)
  Post nerve block | 34 (8.2)

2. Primary Outcome: Peak Pulmonary Arterial Pressure
Description: Measured on exercise cardiopulmonary stress test
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Mmhg
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
Mmhg
  Baseline | 56 (9.2)
  Post nerve block | 47 (10.6)

3. Primary Outcome: Absence of Nerve Block Related Complications
Description: Assessment of orthostasis, gastrointestinal symptoms were observed
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Peak Oxygen Uptake
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mL/min/m2
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
mL/min/m2
  Baseline | 10.5 (2)
  Post nerve block | 9.1 (3)

5. Secondary Outcome: Resting Wedge Pressure
Description: Assessed with right heart cath
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
mmHg
  Baseline | 17.5 (9.5)
  Post nerve block | 14 (1.6)

6. Secondary Outcome: Resting Central Venous Pressure
Description: Assessed with right heart cath
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
mmHg
  Baseline | 9.3 (4.9)
  Post nerve block | 5.8 (2.4)

7. Secondary Outcome: Resting Pulmonary Arterial Pressure
Description: Assessed on right heart catheterization
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
mmHg
  Baseline | 24 (9)
  Post nerve block | 20 (4)

8. Secondary Outcome: Dyspnea - Visual Analog Scale (VAS)
Description: The VAS for dyspnea has a range of 0 to 100, where 0 corresponds to the patient's subjective feeling of "I Can Breathe Normally" and a score of 100 corresponds to "I Can't Breathe At All."
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Splanchnic Nerve Block
Number analyzed (Participants) | 4
units on a scale
  Baseline | 76 (11)
  After nerve block | 81 (21)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Splanchnic Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Splanchnic Nerve Block (N=4)
Pulmonary hemorrhage (Injury, poisoning and procedural complications) | 1 — Pulmonary artery injury with follow up right heart catheterization. Not related to the baseline intervention done a month earlier. Self limited. Patient had no lasting complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT04575428/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT04575428/ICF_001.pdf